CLINICAL TRIAL: NCT01111305
Title: A Randomized, Placebo-controlled, Double-Blind Pilot Study of Single-Dose Humanized Anti-IL5 Antibody (Reslizumab) for the Reduction of Eosinophilia Following Diethylcarbamazine Treatment of Loa Loa Infection
Brief Title: Reslizumab to Prevent Post-treatment Eosinophilia in Loiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-I-0101; 100101 (Other: NIHCC)
Record Dates: First submitted 2010-04-24; First posted 2010-04-27 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2017-10

CONDITIONS: Loiasis
Keywords: Filariasis; Post-Treatment Reactions; Monoclonal Antibody; Loa Loa; Loiasis
MeSH Terms: conditions — Loiasis; Filariasis | interventions — reslizumab; Diethylcarbamazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drug assignment (reslizumab vs. placebo) and eosinophil count
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reslizumab + DEC (Active Comparator): Reslizumab 1 mg/kg iv single dose followed by diethylcarbamazine 9 mg/kg/day po for 21 days
  Interventions: Drug: Reslizumab; Drug: Diethylcarbamazine
- Placebo + DEC (Placebo Comparator): Placebo iv single dose followed by diethylcarbamazine 9 mg/kg/day po for 21 days
  Interventions: Drug: Diethylcarbamazine; Other: Placebo

INTERVENTIONS:
Drug: Reslizumab
  Other Names: Cinqair
  Arms: Reslizumab + DEC
Drug: Diethylcarbamazine
  Other Names: Hetrazan, Banocide
Other: Placebo
  Arms: Placebo + DEC

SUMMARY:
Diethylcarbamazine citrate (DEC) treatment of Loa loa infection is complicated by the development of severe adverse reactions that are correlated with the number of circulating microfilariae in the blood. The cause of these reactions is unknown, but they are accompanied by a dramatic interleukin-5 (IL-5)-dependent increase in eosinophilia and evidence of eosinophil activation. This randomized, placebo-controlled, double-blind pilot study (conducted at the NIH Clinical Center) will assess whether and to what extent the administration of reslizumab (Cinquil ), a humanized monoclonal antibody directed against IL-5, given 3 to 7 days before administration of the anthelminthic drug DEC (at 3 mg/kg 3 times daily for 21 days), prevents the development of eosinophilia in 10 adult subjects with Loa loa infection and 0-5000 microfilariae/mL. Secondary outcomes will include the severity of post-treatment effects, markers of eosinophil activation, and effects of reslizumab on microfilarial clearance.

DETAILED DESCRIPTION:
Background:

Loa loa is a parasitic worm that infects people in West and Central Africa and is spread by the bite of a deerfly. Adult worms (macrofilariae) live under the skin and cause symptoms such as swellings, itching, and hives. Smaller worms (microfilariae) are found in the bloodstream. Diethylcarbamazine (DEC), the recommended medication for Loa loa infection, can produce very serious side effects, especially in people with high numbers of parasites in the blood. Researchers are investigating new treatments for Loa loa that have fewer or less serious side effects. Researchers believe that a certain kind of blood cells called eosinophils, which increase in the blood after DEC treatment, may be one of the causes of the side effects seen with DEC treatment. Reslizumab is a drug that lowers eosinophils in the blood. Giving reslizumab before DEC treatment might prevent the eosinophils from increasing and reduce some of the side effects from DEC.

Objectives:

- To determine whether reslizumab can prevent or reduce the side effects of treatment with DEC for Loa loa infection.

Eligibility:

Screening: Individuals between 18 and 65 years of age who have lived in or traveled to a Loa-endemic region for at least 1 month

Treatment study: Individuals with Loa loa infection and low numbers of parasites in the blood

Design:

This study will last 24 months and will involve several visits to the National Institutes of Health Clinical Center. Participants will be screened with a blood test for Loa loa parasites. Those who have a low number of Loa loa parasites in the blood will be asked to return for a full medical evaluation and the start of the treatment phase. Those who do not have Loa loa parasites in the blood, or those who have a high number of Loa loa parasites in the blood, are not eligible for this study treatment but may be eligible for other parasitic disease studies conducted by the National Institutes of Health.

Participants will have an initial visit with a full physical evaluation, and blood and urine tests (including leukapheresis to provide sufficient numbers of blood cells for testing). Within 1 month of the first visit, participants will have a single infusion of either reslizumab or a placebo. The infusion visit is estimated to last approximately 5 hours. Three to 7 days after the infusion, participants will begin a 21-day course of DEC (taken by mouth) to treat the infection. Participants will stay overnight at the Clinical Center during the first 3 days of treatment with DEC to be monitored for side effects, and will continue to take the DEC at home after the inpatient treatment. A study coordinator will call participants each day to ask about any symptoms or side effects. Participants will be seen for an additional eight outpatient follow-up visits (at days 7, 14, and 28, and months 3, 6, 12, 18, and 24) for evaluation of signs and symptoms of infection.

ELIGIBILITY:
* INCLUSION CRITERIA: (Screening)

A subject will be eligible for participation in the screening portion of this protocol if all of the following criteria apply:

1. Between 18 and 65 years of age
2. Residence in or travel to a Loa-endemic region for greater than 1 month

EXCLUSION CRITERIA: (Screening)

A subject will not be eligible for participation in the screening portion of this study if any of the following conditions apply:

1. Known to be pregnant
2. Known to be HIV-positive

INCLUSION CRITERIA: (Interventional Study)

A subject will be eligible for participation in the interventional portion of the study only if all of the following criteria apply:

1. The subject has documented loiasis with 0-5000 microfilariae/mL blood.
2. The subject agrees to storage of samples for study
3. A female subject is eligible for this study if she is any of the following:

   * Not pregnant or breast-feeding.
   * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are post-menopausal, as defined by no menses in greater than or equal to 1 year)
   * Of childbearing potential but agrees to practice effective contraception* or abstinence for 3 months after administration of the investigational study drug (reslizumab or placebo)

     * NOTE: Acceptable methods of contraception may include one or more of the following: 1) male partner who is sterile prior to the female subject s entry into the study and is the sole sexual partner for the female subject; 2) implants of levonorgestrel; 3) injectable progestogen, an intrauterine device with a documented failure rate of less than 1percent; 4) oral contraceptives; and 5) double barrier methods including diaphragm or condom with a spermicide.

EXCLUSION CRITERIA: (Interventional Study)

A subject will not be eligible to participate in the interventional portion of the study if any of the following conditions are fulfilled at the time of enrollment:

1. The subject tests positive for HIV infection or has any other known immunodeficiency.
2. The subject has a concomitant active infection with Onchocerca volvulus.
3. The subject has used any other investigational agent within the past 30 days.
4. The subject has used immunosuppressive agents (as listed in section 8.1) within the past 30 days.
5. The subject has a history of allergic reaction to any antibody therapy or to DEC.
6. The subject has chronic kidney or liver disease.
7. The subject has any condition that, in the Investigator s opinion, places the subject at undue risk by participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2016-01 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limaye AP, Abrams JS, Silver JE, Ottesen EA, Nutman TB. Regulation of parasite-induced eosinophilia: selectively increased interleukin 5 production in helminth-infected patients. J Exp Med. 1990 Jul 1;172(1):399-402. doi: 10.1084/jem.172.1.399. PMID 2193099
- [Background] Klion AD, Massougbodji A, Sadeler BC, Ottesen EA, Nutman TB. Loiasis in endemic and nonendemic populations: immunologically mediated differences in clinical presentation. J Infect Dis. 1991 Jun;163(6):1318-25. doi: 10.1093/infdis/163.6.1318. PMID 2037798
- [Background] Klion AD, Ottesen EA, Nutman TB. Effectiveness of diethylcarbamazine in treating loiasis acquired by expatriate visitors to endemic regions: long-term follow-up. J Infect Dis. 1994 Mar;169(3):604-10. doi: 10.1093/infdis/169.3.604. PMID 8158033
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-I-0101.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 subjects were enrolled on the screening phase of this protocol, of which 13 had Loa loa infection. Of these 13, 3 were excluded for Loa loa microfilarial loads that were too high, 1 could not comply with the trial time points, and one was lost to followup. This left 8 subjects who were enrolled on the treatment portion of the study.
Groups:
- Reslizumab: Reslizumab
  Diethylcarbamazine
- Placebo: Placebo
  Diethylcarbamazine
Period: Overall Study
Arm/Group | Reslizumab | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reslizumab | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Full Range); unit: years] | 36 [22 to 44] | 29 [20 to 55] | 31.5 [20 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
Loa loa microfilarial level [Geometric Mean (Full Range); unit: mf/mL] | 212 [0 to 2120] | 357 [178 to 810] | 275 [0 to 2120]
Absolute eosinophil count [Geometric Mean (Full Range); unit: cells/microliter] | 1350 [530 to 3130] | 710 [560 to 1590] | 980 [530 to 3130]

OUTCOME MEASURES:

1. Primary Outcome: Peak Eosinophil Count Post-treatment
Description: Peak eosinophil count during the first 7 days of treatment as a percent of the baseline count
Time Frame: during the first 7 days of DEC treatment
Population: Subjects who received diethylcarbamazine treatment
Measure: Geometric Mean (Full Range); unit: percent of baseline eosinophil count
Groups:
- Reslizumab + DEC: Reslizumab 1 mg/kg iv single dose followed by diethylcarbamazine 9 mg/kg/day po for 21 days
  Reslizumab
  Diethylcarbamazine
- Placebo + DEC: Placebo iv single dose followed by diethylcarbamazine 9 mg/kg/day po for 21 days
  Diethylcarbamazine
  Placebo
Arm/Group | Reslizumab + DEC | Placebo + DEC
Number analyzed (Participants) | 4 | 4
percent of baseline eosinophil count | 61 [42.7 to 104] | 245.6 [175 to 372]
Statistical Analysis 1: Comparison: Reslizumab + DEC vs Placebo + DEC; Test type: Equivalence — Equivalence is defined as p≥0.05; p = 0.028, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Frequency of AE's
Description: Adverse events during the first week of DEC treatment
Time Frame: 7 days following initiation of DEC treatment
Population: Subjects who received DEC treatment
Measure: Number; unit: adverse events
Arm/Group | Reslizumab + DEC | Placebo + DEC
Number analyzed (Participants) | 4 | 4
adverse events | 29 | 28

3. Secondary Outcome: Markers of Eosinophil Activation
Description: serum eosinophil granule protein levels on day 7 measured as % baseline
Time Frame: one week
Measure: Geometric Mean (Full Range); unit: % change
Arm/Group | Reslizumab + DEC | Placebo + DEC
Number analyzed (Participants) | 4 | 4
% change
  % day 0 EDN at day 7 | 115 [101 to 132] | 377 [163 to 634]
  % day 0 EPO at day 7 | 138 [92 to 161] | 203 [82 to 344]

4. Secondary Outcome: Proportion of Subjects Who Clear Blood Microfilariae
Time Frame: 3, 7, and 28 days after initiation of treatment with DEC
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  3 days | 2 | 2
  7 days | 4 | 4
  28 days | 4 | 4

ADVERSE EVENTS:
Time Frame: 7 days
Description: A standardized questionnaire was used to record symptoms at every visit. Laboratory assessments were performed at every visit.
Arm/Group | Reslizumab + DEC | Placebo + DEC
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reslizumab + DEC (N=4) | Placebo + DEC (N=4)
Fatigue (General disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Headache (General disorders) | 2 | 2
Calabar swelling (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
LDH increased (Investigations) | 1 | 2
ALT increased (Investigations) | 2 | 1
AST increased (Investigations) | 3 | 2
Bilirubin increased (Investigations) | 1 | 2
CPK increased (Investigations) | 2 | 1
Hematuria (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No